CLINICAL TRIAL: NCT03537248
Title: Clinical Safety and Effectiveness of ASP-57 Multi-Purpose Contact Lens Care Solution Compared to a Marketed Contact Lens Solution
Brief Title: A Safety and Effectiveness Study of a New Multi-Purpose Contact Lens Care Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asepticys LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASP-57-101
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2018-06

CONDITIONS: Contact Lens Wear

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Asepticys investigational ASP-57 Multi-Purpose Solution (Experimental): ASP-57 Multi-Purpose contact lens care solution used as a rub care regimen (Test)
  Interventions: Device: ASP-57
- ReNu® Multiplus Contact Lens Solution (Active Comparator): ReNu® Multiplus Contact Lens Solution used as rub care regimen (Control)
  Interventions: Device: ReNu® Multiplus

INTERVENTIONS:
Device: ASP-57 — an experimental solution for disinfecting, cleaning, conditioning, rinsing, protein removal, ad storing soft contact lenses including silicone hydrogel lenses
  Other Names: Investigational Multi-Purpose Contact Lens Care Solution
  Arms: Asepticys investigational ASP-57 Multi-Purpose Solution
Device: ReNu® Multiplus — a multi-purpose solution for disinfecting, cleaning, conditioning, rinsing, protein removal, ad storing soft contact lenses including silicone hydrogel lenses
  Arms: ReNu® Multiplus Contact Lens Solution

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of ASP-57 Multi-Purpose contact lens solution (Test) compared to ReNu® Multiplus Contact Lens Solution (Control) when used by habitual contact lens wearers to bilaterally clean and disinfect their contact lenses for approximately 3 months (12 weeks).

DETAILED DESCRIPTION:
Approximately 330 subjects (660 eyes) will be enrolled in this 3 month (12 week) controlled, parallel group, masked, randomized study at approximately 15 investigative sites in the United States. Subjects will be randomized 2:1 to receive either Asepticys ASP-57 Multi-Purpose Solution or ReNu® Multiplus Contact Lens Solution (Control) respectively. Both Test and Control solution will be used with a rub care regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age ≥ 18 years on the date of informed consent.
2. All subjects must provide signed written consent prior to participation in any study related procedures.
3. Successful history of wear of the one of the following lens types (toric and multifocal lenses of the specified lens type are allowed) in both eyes during the past 3 months, and history of at least 5 consecutive days of successful daily wear in both eyes prior to Visit 1:

   * All Bausch & Lomb PureVision lens types
   * All Alcon Air Optix lens types
   * All CooperVision Biofinity lens types
   * All Vistakon Acuvue Oasys lens types
   * Any conventional hydrogel Group IV lens
4. Vision correctable through spherocylindrical refraction to 32 letters (0.3 logMAR) or better (distance, high contrast) in each eye.
5. Clear central corneas and free of any anterior segment disorders
6. Habitual use of a Multi-Purpose Solution for cleaning, disinfecting, and storage of lenses.
7. Lens correction in both eyes is required and the same brand of lens is worn in each eye.
8. Agree to wear study lenses in both eyes on a daily wear basis, with lenses removed every night (not slept in) throughout the study period and no lens or pair of lenses worn for longer than 2 weeks.
9. Able and willing to comply with all care regimen and follow-up study procedures.

Exclusion Criteria:

1. Females of childbearing potential (not surgically sterilized or postmenopausal) if any one of the following conditions are met:

   * currently pregnant,
   * plan to become pregnant during the study,
   * are breast-feeding.
2. Wear of gas permeable contact lenses within the last 30 days.
3. Wear of polymethylmethacrylate lenses within the last 3 months.
4. No topical ocular prescription medications may be administered during the study period. Ongoing use of non-preserved artificial tears up to 4 times daily (with no changes in frequency or brand) is allowed. Ongoing use of the rewetting drop the subject customarily uses (with no switch in brand or type) is also permitted during the study period.
5. Current systemic disease affecting ocular health or use of topical or systemic medications that, in the Investigator's opinion, could affect ocular physiology or lens performance.
6. Ocular astigmatism of 2.00 D or greater in either eye based on the contact lens prescription.
7. Grade 2 or greater finding on any slit-lamp scale and/or corneal infiltrates of any grade during slit-lamp examination at Screening.
8. Any finding during slit-lamp examination that, in the Investigator's opinion, interferes with contact lens wear.
9. Scar or neovascularization within the central 4 millimeters (mm) of the cornea. Minor peripheral corneal scarring (that does not extend into the central zone) is permitted, if in the Investigator's judgment, it does not interfere with contact lens wear.
10. Aphakia.
11. Amblyopia.
12. History of any corneal surgery.
13. Allergy to any component of the study solutions.
14. Participation in any clinical study within the 2 weeks prior to entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Slit Lamp Findings | 3 months
  Statistical non-inferiority with respect to the proportion of eyes with any slit-lamp findings greater than Grade 2 at any visit between the test and control solutions
Visual Acuity | 3 months
  Statistical non-inferiority with respect to the proportion of subjects with greater than 2-line worsening in visual acuity in any eye at any visit between the test and control solutions

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Lakeside Vision Center, Irvine, California
  - Complete Family Vision Care, San Diego, California
  - Sabal Eye Care, Longwood, Florida
  - Maitland Vision Center, Maitland, Florida
  - Vision Health Institute, Orlando, Florida
  - Eye Care Associates, Bloomington, Illinois
  - Kannarr Eye Care, Pittsburg, Kansas
  - Heart of America Eye Care, Shawnee Mission, Kansas
  - Seidenberg Protzko Eye Associates, Havre de Grace, Maryland
  - Insight Eyecare, Warrensburg, Missouri
  - Drs Quinn, Foster & Associates, Athens, Ohio
  - West Bay Eye, Warwick, Rhode Island
  - Optometry Group, Memphis, Tennessee
  - Optique Eyecare, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No